CLINICAL TRIAL: NCT03259516
Title: Pilot Open-label Trial of Nivolumab Combined With Chemotherapy in Refractory Myelodysplastic Syndromes.
Brief Title: Nivolumab With Chemotherapy in Refractory MDS
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Slow recruitment rate
Sponsor: St. Petersburg State Pavlov Medical University (Other)
Responsible Party: Principal Investigator, Ivan S Moiseev, Vice-director for science, R.M. Gorbacheva memorial institute, St. Petersburg State Pavlov Medical University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18/17-n
Record Dates: First submitted 2017-08-22; First posted 2017-08-23 (Actual); Last update posted 2019-04-05 (Actual); Status verified 2019-04

CONDITIONS: Myelodysplastic Syndromes
Keywords: myelodysplastic syndrome; nivolumab; 5-azacitidine; cytarabine; melphalan; all-trans retinoic acid; lymphodepletion
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — Nivolumab; Azacitidine; fludarabine; Cyclophosphamide; Cytarabine; Tretinoin; Sildenafil Citrate; Melphalan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Nivo + FC (Experimental): Nivolumab 1 mg/kg days 1,15 iv q28days Fludarabine 25 mg/m2 days 1-3 iv q28days Cyclophosphamide 300 mg/m2 days 1-3 iv q28days
  Interventions: Drug: Nivolumab; Drug: Fludarabine; Drug: Cyclophosphamide
- Nivo + LDAC + ATRA (Experimental): Nivolumab 1 mg/kg days 1,15 iv q28days Cytarabine 10 mg/m2 bid days 1-10 sc q28days All-trans retinoic acid (ATRA) 45 mg/m2 po qd
  Interventions: Drug: Nivolumab; Drug: Cytarabine; Drug: all trans retinoic acid
- Nivo + LDAC + Sildenafil (Experimental): Nivolumab 1 mg/kg days 1,15 iv q28days Cytarabine 10 mg/m2 bid days 1-10 sc q28days Sildenafil 20 mg tid
  Interventions: Drug: Nivolumab; Drug: Cytarabine; Drug: Sildenafil
- Nivo + Melphalan (Experimental): Nivolumab 1 mg/kg days 1,15 iv q28days Melphalan 2 mg qd days 1-10 q28days
  Interventions: Drug: Nivolumab; Drug: Melphalan
- Nivo + 5-aza (Experimental): Nivolumab 1 mg/kg days 1,15 iv q28days 5-azacitidine 75 mg/m2 days 1-7 q28days
  Interventions: Drug: Nivolumab; Drug: Azacitidine

INTERVENTIONS:
Drug: Nivolumab — 1 mg/kg by vein on Days 1 and 15 of a 28 day cycle
  Other Names: Opdivo
Drug: Azacitidine — 75 mg/m2 subcutaneously on Days 1-7 of a 28 day cycle
  Other Names: 5-azacitidine; Vidaza
  Arms: Nivo + 5-aza
Drug: Fludarabine — 25 mg/m2 by vein on Days 1, 2 and 3 of a 28 day cycle. Dose reduction to 15 mg/m2 is permitted in cases of grade 4 hematological toxicity after first cycle.
  Arms: Nivo + FC
Drug: Cyclophosphamide — 300 mg/m2 by vein on Days 1, 2 and 3 of a 28 day cycle.
  Arms: Nivo + FC
Drug: Cytarabine — 10 mg/m2 subcutaneously two times a day on Days 1-10 of a 28 day cycle
  Other Names: Ara-C, LDAC
  Arms: Nivo + LDAC + ATRA; Nivo + LDAC + Sildenafil
Drug: all trans retinoic acid — 45 mg/m2 per os daily during the whole course of treatment
  Other Names: ATRA
  Arms: Nivo + LDAC + ATRA
Drug: Sildenafil — 20 mg per os three times a day during the whole course of treatment
  Arms: Nivo + LDAC + Sildenafil
Drug: Melphalan — 2 mg per os daily during the whole course of treatment
  Arms: Nivo + Melphalan

SUMMARY:
There is evidence of involvement of checkpoint pathways, including PD-1, in the pathogenesis and resistance of myelodysplastic syndrome (MDS). However monotherapy with checkpoint inhibitors was ineffective in a number of studies, indicating the presence of several mechanisms of resistance. This pilot study evaluates the safety and preliminary efficacy of nivolumab combination with currently existing treatments in MDS patients who failed at least one line of therapy. The study evaluates if there is a combination which induces objective responses.

ELIGIBILITY:
Inclusion Criteria:

* Patients with myelodysplastic syndrome (MDS) (up to 20% blasts) of any risk. Patients with lower risk MDS (low and int-1 by IPSS) should have failed prior non-hypomethylating agent therapy (ie growth factors or lenalidomide). Patients with higher risk MDS (int-2 or high by IPSS) should have failed prior at least one therapy with a hypomethylating agent or Ara-C.
* Age 18 years or older.
* No severe organ dysfunction: creatinine <=2.5 x ULN; serum bilirubin <=2.5 x ULN; AST and ALT <=5 x ULN.
* Karnofsky index >=70%
* Females of childbearing potential must have a negative serum or urine beta human chorionic gonadotrophin (beta-hCG) pregnancy test result within 24 hours prior to the first dose of treatment and must agree to use an effective contraception to avoid pregnancy for 24 weeks
* Males who have partners of childbearing potential must agree to use an effective contraceptive method during the study and for 24 weeks after the last dose of nivolumab.

Exclusion Criteria:

* Another malignancy requiring treatment at the time of inclusion
* History of interstitial lung disease or pneumonitis
* Patients with any other known concurrent severe and/or uncontrolled medical condition (e.g. uncontrolled diabetes; cardiovascular disease including congestive heart failure NYHA Class III or IV, myocardial infarction within 6 months, and poorly controlled hypertension; chronic renal failure; or active uncontrolled infection) which, in the opinion of the investigator could compromise participation in the study
* Active, known or suspected autoimmune disease requiring treatment at the time of inclusion
* Pregnancy or breastfeeding
* Patients unwilling or unable to comply with the protocol
* Somatic or psychiatric disorder making the patient unable to sign informed consent
* Prior treatment with anti-PD-1, anti-PD-L1, or anti-CTLA4 therapy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2017-05-25 (Actual); Primary Completion 2018-12-25 (Actual); Study Completion 2018-12-25 (Actual)

PRIMARY OUTCOMES:
Overall response rate | 6 months
  Overall response rate (ORR) defined as complete response plus partial response (CR + PR) and hematological improvement (HI). MDS International Working Group criteria will be used to assess response.

SECONDARY OUTCOMES:
Treatment-related adverse events as assessed by CTCAE v4.03 | 6 months
  Toxicity parameters based on NCI CTCAE 4.03 grades: hematological toxicity (CBC), hepatotoxicity (liver function tests), nephrotoxicity (creatinine), neurotoxicity (attending physician assessment), fatigue (attending physician assessment), rash (attending physician assessment), colitis (attending physician assessment), pneumonitis (attending physician assessment), autoimmune disorders (level of hormones, presence of autoimmune antibodies, attending physician assessment).
Infectious complications | 6 months
  Incidence of severe bacterial, fungal and viral infections incidence based on laboratory confirmation and attending physician assessment

CONTACTS AND LOCATIONS:
Locations (1):
- First Pavlov State Medical University of St. Petersburg, Saint Petersburg, Russia

IPD SHARING:
Plan to Share IPD: Undecided